CLINICAL TRIAL: NCT05206513
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, and Tolerability of Valbenazine for the Treatment of Dyskinesia Due to Cerebral Palsy
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of Valbenazine for the Treatment of Dyskinesia Due to Cerebral Palsy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-DCP3018; EUCT (Other: 2022-502713-29-00)
Record Dates: First submitted 2022-01-10; First posted 2022-01-25 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Dyskinesia; Cerebral Palsy
Keywords: Cerebral Palsy; Vesicular monoamine transporter 2 (VMAT2) inhibitor; Dyskinesia; Neurocrine; Valbenazine; NBI-98854; Dystonia; Chorea; Athetosis; Athetoid cerebral palsy; Choreoathetosis
MeSH Terms: conditions — Dyskinesias; Cerebral Palsy; Dystonia; Chorea; Athetosis | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo dosed for 14 weeks (double-blind treatment period) followed by open-label valbenazine treatment.
  Participants may opt to enter an open-label valbenazine treatment extension phase.
  Interventions: Drug: Placebo; Drug: Valbenazine
- Valbenazine (Experimental): Valbenazine dosed for 14 weeks (double-blind treatment period) followed by open-label valbenazine treatment.
  Participants may opt to enter an open-label valbenazine treatment extension phase.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Placebo — Capsule, administered once daily orally or via gastrostomy/gastrojejunostomy tube
  Arms: Placebo
Drug: Valbenazine — Capsule, administered once daily orally or via gastrostomy/gastrojejunostomy tube
  Other Names: NBI-98854

SUMMARY:
The primary objective of this study is to evaluate the efficacy of valbenazine versus placebo on improving chorea in pediatric and adult participants who have dyskinesia due to cerebral palsy (DCP) with choreiform movements.

ELIGIBILITY:
Key Inclusion Criteria:

1. Medically confirmed diagnosis of DCP (that is, a hyperkinetic movement disorder due to cerebral palsy [CP]) with choreiform movements.
2. Medical conditions are stable and expected to remain stable throughout the study.

Key Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Are pregnant or breastfeeding.
2. Have a clinical diagnosis or history of dyskinesia due to condition other than CP.
3. Have inability to swallow soft foods, unless medications can be administered via gastrostomy/gastrojejunostomy tube.
4. Have any suicidal behavior or suicidal ideation in the year prior to screening or on Day 1.
5. Is a substance abuser of any compound.
6. Known history of long QT syndrome or cardiac tachyarrhythmia, or clinically significant electrocardiogram (ECG) abnormalities.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Total Maximal Chorea (TMC) Score of the Unified Huntington Disease Rating Scale (UHDRS) from Baseline to the Average of the Week 12 and Week 14 assessments | Baseline, Week 12 and Week 14

SECONDARY OUTCOMES:
Change in the Clinical Global Impression of Severity (CGI-S) Score from Baseline to Week 14 | Baseline, Week 14
Change in the Movement Disorders - Childhood Rating Scale (MD-CRS) Part I Score from Baseline to the Average of the Week 12 and Week 14 Assessments | Baseline, Week 12 and Week 14
Change in the Total Maximal Dystonia (TMD) Score of the UHDRS from Baseline to the Average of the Week 12 and Week 14 Assessments | Baseline, Week 12 and Week 14
Patient Global Impression of Improvement (PGI-I) Score at Week 14 | Week 14
Caregiver Global Impression of Improvement (CaGI-I) Score at Week 14 | Week 14
Clinical Global Impression of Improvement (CGI-I) Score at Week 14 | Week 14
Goal Attainment Score at Week 14 Using the Goal Attainment Scale (GAS) | Week 14
Change in Pain Assessment from Baseline to Week 14 Using the Faces Pain Scale-Revised (FPS-R) | Baseline, Week 14
Change in the UHDRS Total Motor Score (TMS) from Baseline to the Average of the Week 12 and Week 14 Assessments | Baseline, Week 12 and Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (35):
- United States (19):
  - Neurocrine Clinical Site, San Diego, California
  - Neurocrine Clinical Site, Aurora, Colorado
  - Neurocrine Clinical Site, Stamford, Connecticut
  - Neurocrine Clinical Site, Gulf Breeze, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Orlando, Florida
  - Neurocrine Clinical Site, Chicago, Illinois
  - Neurocrine Clinical Site, Baltimore, Maryland
  - Neurocrine Clinical Site, Boston, Massachusetts
  - Neurocrine Clinical Site, Farmington Hills, Michigan
  - Neurocrine Clinical Site, Saint Paul, Minnesota
  - Neurocrine Clinical Site, New York, New York
  - Neurocrine Clinical Site, Cincinnati, Ohio
  - Neurocrine Clinical Site, Columbus, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, Portland, Oregon
  - Neurocrine Clinical Site, Dallas, Texas
  - Neurocrine Clinical Site, Fort Worth, Texas
  - Neurocrine Clinical Site, Houston, Texas
- Neurocrine Clinical Site, Buenos Aires, Argentina
- Neurocrine Clinical Site, Brussels, Belgium
- Brazil (3):
  - Neurocrine Clinical Site, Brasília
  - Neurocrine Clinical Site, Curitiba
  - Neurocrine Clinical Site, Porto Alegre
- Neurocrine Clinical Site, Ẕerifin, Israel
- Italy (2):
  - Neurocrine Clinical Site, Calambrone
  - Neurocrine Clinical Site, Milan
- Neurocrine Clinical Site, Aguascalientes, Mexico
- Poland (3):
  - Neurocrine Clinical Site, Gdansk
  - Neurocrine Clinical Site, Krakow
  - Neurocrine Clinical Site, Oświęcim
- Portugal (2):
  - Neurocrine Clinical Site, Lisbon
  - Neurocrine Clinical Site, Porto
- Spain (2):
  - Neurocrine Clinical Site, Barcelona
  - Neurocrine Clinical Site, Madrid

IPD SHARING:
Plan to Share IPD: No